CLINICAL TRIAL: NCT02344641
Title: Efficacy and Mechanism of Exenatide on Improving Heart Function in Type 2 Diabetes With Heart Failure Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, YanYan Chen, Director，endocrinology and cardiology centre, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISSEXEN0054
Record Dates: First submitted 2015-01-13; First posted 2015-01-26 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes Mellitus; Heart Failure
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exenatide (Experimental): exenatide group receive exenatide (5μg, subcutaneous injection, Bid）
  Interventions: Drug: Exenatide
- control group (No Intervention): control group do not receive exenatide

INTERVENTIONS:
Drug: Exenatide
  Arms: Exenatide

SUMMARY:
The study evaluates the efficacy of heart function improvements in type 2 diabetes and heart failure patients with exenatide, and also investigates the mechanisms of exenatide improving heart function.

DETAILED DESCRIPTION:
The study enrolls 234 patients with type 2 diabetes and heart failure. The patients have an New York Heart Association (NYHA) functional class of II to IV, are randomly assigned to 2 groups. One group use exenatide , the other group is control group and each group has 117 patients. At the baseline, the 3rd day, the 28th day patients are required to complete the heart failure examination: plasma N-terminal pro-B-type natriuretic peptide(NT-proBNP), 6-min walking distance, echocardiographic measures, patient quality of life(MLHFQ). At the end of 4-week follow-up, we evaluate the efficacy of heart function improvements after treatment with exenatide and also investigate the mechanisms of exenatide improving heart function .

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed Type 2 diabetes mellitus
2. HbA1c 7%-10% and Fasting plasma glucose(FBG) <10mmol/L
3. Age 18-65 years
4. NT-proBNP level≥ 450 pg/ml
5. Left ventricular ejection fraction (LVEF)<40%

Exclusion Criteria:

1. Uncorrected primary vascular disease
2. congenital heart disease
3. Left ventricular outflow obstruction
4. Myocarditis
5. Aneurysm
6. uncontrolled severe arrhythmia
7. cardiogenic shock
8. unstable angina, or acute myocardial infarction
9. Severe primary hepatic, renal, or hematologic disease
10. Cr>194.5 mmol/l or K+>5.5 mmol/l
11. Systolic blood pressure (SBP) ≥180mm Hg or diastolic blood pressure (DBP) ≥110mm Hg
12. Alanine aminotransferase (ALT) >3 times the upper normal limit
13. Patients were likely to undergo coronary artery bypass graft surgery during the following 4 weeks
14. Patients had undergone or were likely to undergo cardiac resynchronization therapy
15. Pregnant or lactating known
16. Suspected to be allergic to the study drugs
17. Use dipeptidyl peptidase-4 (DPP-4) or glucagon-like peptide-1 (GLP-1) drug in 3 months
18. Hyperthyroidism and Hypothyroidism
19. Tumor
20. Received another investigational drug within 30 days prior to randomization
21. Severe mental health condition or other uncontrolled systemic disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The change in plasma NT-proBNP level after using exenatide for 4 weeks | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: YanYan Chen, MD, Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Disease